CLINICAL TRIAL: NCT02050919
Title: A Phase II Study of Sorafenib With Chemotherapy, Radiation, and Surgery for High-Risk Soft Tissue Sarcomas
Brief Title: Sorafenib Tosylate, Combination Chemotherapy, Radiation Therapy, and Surgery in Treating Patients With High-Risk Stage IIB-IV Soft Tissue Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Bayer (Industry); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Christopher Ryan, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00009464; NCI-2013-02414 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IRB00009464 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2014-01-29; First posted 2014-01-31 (Estimated); Results first posted 2020-06-11 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-02

CONDITIONS: Pleomorphic Rhabdomyosarcoma; Stage IIB Adult Soft Tissue Sarcoma AJCC v7; Stage III Adult Soft Tissue Sarcoma AJCC v7; Stage IV Adult Soft Tissue Sarcoma AJCC v7
MeSH Terms: conditions — Sarcoma | interventions — Epirubicin; Ifosfamide; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (sorafenib, chemotherapy, radiation, surgery) (Experimental): Patients receive sorafenib tosylate PO QD on days 1-71 and 85-155, epirubicin hydrochloride IV over 3-5 minutes, and ifosfamide IV over 90 minutes on days 15-17, 36-38 (ifosfamide only), 57-59, 99-101, 120-122, and 141-143. Patients undergo EBRT on days 36-45 and surgical resection on day 78. Patients with positive margins, undergo EBRT boost on days 91-98.
  Interventions: Drug: Epirubicin Hydrochloride; Radiation: External Beam Radiation Therapy; Drug: Ifosfamide; Other: Laboratory Biomarker Analysis; Drug: Sorafenib Tosylate; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Drug: Epirubicin Hydrochloride — Given IV
  Other Names: Ellence; IMI-28; Pharmorubicin PFS
Radiation: External Beam Radiation Therapy — Undergo EBRT
  Other Names: Definitive Radiation Therapy; EBRT; External Beam Radiotherapy; External Beam RT; external radiation; External Radiation Therapy; external-beam radiation
Drug: Ifosfamide — Given IV
  Other Names: Asta Z 4942; Asta Z-4942; Cyfos; Holoxan; Holoxane; Ifex; IFO; IFO-Cell; Ifolem; Ifomida; Ifomide; Ifosfamidum; Ifoxan; IFX; Iphosphamid; Iphosphamide; Iso-Endoxan; Isoendoxan; Isophosphamide; Mitoxana; MJF 9325; MJF-9325; Naxamide; Seromida; Tronoxal; Z 4942; Z-4942
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Sorafenib Tosylate — Given PO
  Other Names: BAY 43-9006 Tosylate; BAY 54-9085; Nexavar; sorafenib
Procedure: Therapeutic Conventional Surgery — Undergo surgical resection

SUMMARY:
This phase II trial studies how well sorafenib tosylate, combination chemotherapy, radiation therapy, and surgery work in treating patients with high-risk stage IIB-IV soft tissue sarcoma. Sorafenib tosylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as epirubicin hydrochloride and ifosfamide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Radiation therapy uses high energy x rays to kill tumor cells. Giving sorafenib tosylate, combination chemotherapy, radiation therapy, and surgery may be an effective treatment for soft tissue sarcoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the pathologic response rate (>= 95% necrosis) after preoperative treatment with sorafenib (sorafenib tosylate), epirubicin (epirubicin hydrochloride), ifosfamide, and hypofractionated radiation for high risk soft tissue sarcomas of the extremities or body wall.

SECONDARY OBJECTIVES:

I. To further characterize the safety of sorafenib plus chemoradiotherapy, including wound complication rate.

II. To estimate time-to-event rates, including overall survival, overall disease-free survival, distant disease-free survival, and local disease-free survival in patients with high risk soft tissue sarcomas of the extremities or body wall treated with preoperative sorafenib plus chemoradiotherapy and postoperative sorafenib plus chemotherapy.

OUTLINE:

Patients receive sorafenib tosylate orally (PO) once daily (QD) on days 1-71 and 85-155, epirubicin hydrochloride intravenously (IV) over 3-5 minutes, and ifosfamide IV over 90 minutes on days 15-17, 36-38 (ifosfamide only), 57-59, 99-101, 120-122, and 141-143. Patients undergo external beam radiation therapy (EBRT) on days 36-45 and surgical resection on day 78. Patients with positive margins, undergo EBRT boost on days 91-98.

After completion of study treatment, patients are followed up every 4 months for 2 years, every 6 months for 1 year, and then yearly for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, soft-tissue sarcoma: excluding rhabdomyosarcoma (pleomorphic rhabdomyosarcoma patients are eligible), Ewing's, primitive neuroectodermal tumor (PNET), osteosarcoma, or gastrointestinal stromal tumor
* American Joint Committee on Cancer (AJCC) (7th edition) stage IIb, III, or IV patients planned for resection of the primary tumor

  * > 5 cm in greatest dimension
  * Intermediate or high-grade
  * Superficial or deep
* Sarcoma located on upper (includes shoulder) or lower (includes hip) extremities or on body wall
* Intermediate or high-grade: grades 2 or 3 on scale of 1-3
* Left ventricular ejection fraction (LVEF) >= 50%
* Absolute neutrophil count (ANC) >= 1500/uL
* Hemoglobin (Hgb) >= 9.0 g/dL
* Platelets >= 100,000/uL
* Creatinine =< 1.5 x upper limit of normal (ULN)
* Bilirubin =< 1.5 mg/dL
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 1.5 x ULN
* International normalized ratio (INR) < 1.5 or a prothrombin time (PT)/partial thromboplastin time (PTT) within normal limits; patients receiving anti-coagulation treatment with an agent such as warfarin or heparin may be allowed to participate; for patients on warfarin, the INR should be measured prior to initiation of sorafenib and monitored at least weekly, or as defined by the local standard of care, until INR is stable
* No prior chemotherapy, radiation, or biotherapy
* No major surgery within 4 weeks prior to study entry
* No contraindications to limb-sparing surgery; patient should be evaluated by a surgeon who specializes in sarcoma resections prior to study enrollment to ensure patient (pt) is a candidate for limb-sparing surgery
* No severe peripheral vascular disease
* Adequate contraception must be used and patients must not be pregnant or breastfeeding; women of childbearing potential and men must agree to use adequate contraception (barrier method of birth control) prior to study entry and for the duration of study participation; men and women should use adequate birth control for at least thirty days after the last administration of sorafenib
* Women of childbearing potential must have negative serum pregnancy test performed within 7-days prior to registration
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1
* Patient must sign a study-specific consent form prior to registration
* Ability to understand and the willingness to sign a written informed consent; a signed informed consent must be obtained prior to any study specific procedures

Exclusion Criteria:

* Patients with known brain metastases; patients with neurological symptoms must undergo a computed tomography (CT) scan/magnetic resonance imaging (MRI) of the brain to exclude brain metastases
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active serious infection > Common Terminology Criteria for Adverse Events (CTCAE) grade 2, symptomatic congestive heart failure, unstable angina pectoris, cardiac ventricular arrhythmia requiring anti-arrhythmic therapy, or psychiatric illness/social situations that would limit compliance with study requirements; patients must not have unstable angina (angina symptoms at rest) or new onset angina (began within the last 3 months) or myocardial infarction within the past 6 months
* Uncontrolled hypertension defined as systolic blood pressure > 150 mmHg or diastolic pressure > 90 mmHg, despite optimal medical management
* Known human immunodeficiency virus (HIV) infection or chronic hepatitis B or C
* Thrombolic or embolic events such as a cerebrovascular accident including transient ischemic attacks within the past 6 months
* Pulmonary hemorrhage/bleeding event >= CTCAE grade 2 within 4 weeks of first dose of study drug
* Any other hemorrhage/bleeding event >= CTCAE grade 3 within 4 weeks of first dose of study drug
* Serious non-healing wound, ulcer, or bone fracture
* Evidence or history of bleeding diathesis or coagulopathy
* Major surgery or significant traumatic injury within 4 weeks of first study drug
* Use of strong cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) inducers
* Known or suspected allergy to sorafenib or any agent given in the course of this trial
* Any condition that impairs patient's ability to swallow whole pills
* Any malabsorption problem
* Pregnant or lactating women are excluded from this study
* Patients with a "currently active" second malignancy other than non-melanoma skin cancers are not to be registered; patients are not considered to have a "currently active" malignancy if they have completed therapy and considered by their physician to be at less than 30% risk of relapse
* Any uncontrolled thyroid disease
* Requirement for hemodialysis or peritoneal dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-12-03 (Actual); Primary Completion 2018-05-07 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Ryan, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

REFERENCES:
- [Derived] Vatner R, James CD, Sathiaseelan V, Bondra KM, Kalapurakal JA, Houghton PJ. Radiation therapy and molecular-targeted agents in preclinical testing for immunotherapy, brain tumors, and sarcomas: Opportunities and challenges. Pediatr Blood Cancer. 2021 May;68 Suppl 2:e28439. doi: 10.1002/pbc.28439. Epub 2020 Aug 22. PMID 32827353

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Sorafenib, Chemotherapy, Radiation, Surgery)
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Sorafenib, Chemotherapy, Radiation, Surgery)
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 18
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Response Rate, Defined as the Percentage of Participants With Greater Than or Equal to 95% Necrosis.
Description: Descriptive statistical analysis will be conducted. The proportion with 95% confidence interval will be summarized.
Time Frame: Assessed at surgical resection
Measure: Number (95% Confidence Interval); unit: % of participants
Arm/Group | Treatment (Sorafenib, Chemotherapy, Radiation, Surgery)
Number analyzed (Participants) | 20
% of participants | 20 [5.7 to 43.7]

2. Secondary Outcome: Number of Grade 3-4 Adverse Events
Description: Measured as the number of Grade 3-4 Adverse Events, graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.0
Time Frame: Up to 5 years
Measure: Number; unit: Grade 3-4 Adverse Events
Arm/Group | Treatment (Sorafenib, Chemotherapy, Radiation, Surgery)
Number analyzed (Participants) | 20
Grade 3-4 Adverse Events | 86

3. Secondary Outcome: Number of Participants With Wound Complications
Description: Wound complication rate, including 1) any secondary operation for wound repair, or 2) wound management without secondary operation including invasive procedures without general or regional anesthesia, readmission for wound care, or persistent deep packing for 120 days or longer.
Time Frame: At least 120 days
Population: Patients who had surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Sorafenib, Chemotherapy, Radiation, Surgery)
Number analyzed (Participants) | 20
Participants | 10

4. Secondary Outcome: Overall Survival at 2 Years
Description: Percentage of patients alive at 2 years, Method of Kaplan-Meier used.
Time Frame: Time from registration until death from any cause
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment (Sorafenib, Chemotherapy, Radiation, Surgery)
Number analyzed (Participants) | 20
percentage of patients | 82 [54 to 94]

5. Secondary Outcome: Overall Disease-free Survival (Stage IIB-III Patients)
Description: Time from surgical resection to local recurrence, distant metastatic disease or death, subjects with stage IV disease excluded. Method of Kaplan-Meier \used.
Time Frame: Time from surgical resection to local recurrence, distant metastatic disease, or death, whichever occurs first, assessed up to 2 years
Population: 15 of the 20 patients enrolled on the trial were evaluable for DFS. Four patients were metastatic at baseline, and 1 developed metastatic disease during preoperative treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Sorafenib, Chemotherapy, Radiation, Surgery)
Number analyzed (Participants) | 15
Months | 13.3 [6 to NA] — There were not sufficient events to define the upper limit of the confidence interval.

6. Secondary Outcome: Distant Disease-free Survival (Stage IIB-III Patients)
Description: Time from registration to development of distant metastatic disease or death, subjects with stage IV disease excluded. Method of Kaplan-Meier used.
Time Frame: Time from registration until development of distant metastatic disease or death, whichever occurs first, assessed up to 2 years
Population: Four patients were metastatic at baseline, and thus excluded from the distant disease-free survival evaluation.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Sorafenib, Chemotherapy, Radiation, Surgery)
Number analyzed (Participants) | 16
Months | 16.4 [8.9 to NA] — There were not sufficient events to define the upper limit of the confidence interval.

7. Secondary Outcome: Number of Participants With Local Recurrence
Description: Number of patients with local recurrence after surgical resection of the primary tumor
Time Frame: Time from surgical resection until primary analysis ( Median follow-up for local recurrence 17.11 months, range 6.18 - 42.8 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Sorafenib, Chemotherapy, Radiation, Surgery)
Number analyzed (Participants) | 16
Participants | 0

ADVERSE EVENTS:
Time Frame: Toxicity measure through follow up, every 4 months until patient death or withdrawal, a median of 34.5 months.
Description: Adverse events will be using the NCI Common Toxicity Criteria for Adverse Events v4.0. Assessment of study drug attribution will be made by an Investigator. Acute and long-term radiation toxicity will be assessed for the following CTCAE categories: 1) Injury, poisoning and procedural complications: Dermatitis radiation 2) Musculoskeletal and connective tissue disorders: Fibrosis 3) other appropriate Musculoskeletal and connective tissue disorders AEs appropriate to limb function.
Arm/Group | Treatment (Sorafenib, Chemotherapy, Radiation, Surgery)
All-Cause Mortality (participants affected / at risk) | 5/20
Serious Adverse Events (participants affected / at risk) | 18/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Sorafenib, Chemotherapy, Radiation, Surgery) (N=20)
Catheter Related infection (Infections and infestations) | 1
Constipation (Gastrointestinal disorders) | 1
Delirium (Psychiatric disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Encephalopathy (Nervous system disorders) | 3
enterocolitis infectious (Infections and infestations) | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 12
Hypokalemia (Metabolism and nutrition disorders) | 1
Lymphocyte count decreased (Investigations) | 1
Neutrophil Count decreased (Investigations) | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Platelet Count Decreased (Investigations) | 2
Sepsis (Infections and infestations) | 3
Soft tissue infection (Infections and infestations) | 1
syncope (Nervous system disorders) | 1
wound dehiscence (Injury, poisoning and procedural complications) | 1
wound infection (Infections and infestations) | 7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Sorafenib, Chemotherapy, Radiation, Surgery) (N=20)
Abdominal Pain (Gastrointestinal disorders) | 1
Activated partial thromboplastin time prolonged (Investigations) | 1
Acute Kidney Injury (Renal and urinary disorders) | 2
akathisia (Nervous system disorders) | 1
Alanine aminotransferase increased (Investigations) | 8
Alkaline phosphatase increased (Investigations) | 8
alopecia (Skin and subcutaneous tissue disorders) | 2
anal fistula (Gastrointestinal disorders) | 1
Anemia (Blood and lymphatic system disorders) | 19
anorectal infection (Infections and infestations) | 1
anorexia (Metabolism and nutrition disorders) | 6
anxiety (Psychiatric disorders) | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 2
Aspartate aminotransferase Increased (Investigations) | 10
Atrial flutter (Cardiac disorders) | 1
Bloating (Gastrointestinal disorders) | 1
Blood bilirubin increased (Investigations) | 5
blurred vision (Eye disorders) | 2
bone pain (Musculoskeletal and connective tissue disorders) | 1
Burn (Injury, poisoning and procedural complications) | 1
Catheter Related Infection (Infections and infestations) | 1
Chills (General disorders) | 1
Confusion (Psychiatric disorders) | 1
Constipation (Gastrointestinal disorders) | 8
cough (Respiratory, thoracic and mediastinal disorders) | 2
Creatinine increased (Investigations) | 6
dehydration (Metabolism and nutrition disorders) | 3
Dermatitis radiation (Injury, poisoning and procedural complications) | 6
Diarrhea (Gastrointestinal disorders) | 8
Dizziness (Nervous system disorders) | 2
Dry mouth (Gastrointestinal disorders) | 1
dry skin (Skin and subcutaneous tissue disorders) | 2
Dysgeusia (Nervous system disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Edema limbs (General disorders) | 3
Ejection fraction decreased (Investigations) | 1
encephalopathy (Nervous system disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Fatigue (General disorders) | 10
Febrile Neutropenia (Blood and lymphatic system disorders) | 1
fever (General disorders) | 1
flushing (Vascular disorders) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4
Headache (Nervous system disorders) | 1
Hematuria (Renal and urinary disorders) | 1
hemorrhoids (Gastrointestinal disorders) | 2
hiccups (Respiratory, thoracic and mediastinal disorders) | 2
Hot flashes (Vascular disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 11
hyperkalemia (Metabolism and nutrition disorders) | 2
hypermagnesemia (Metabolism and nutrition disorders) | 2
Hypernatremia (Metabolism and nutrition disorders) | 3
Hypertension (Vascular disorders) | 8
Hypoalbuminemia (Metabolism and nutrition disorders) | 16
hypocalcemia (Metabolism and nutrition disorders) | 12
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 11
Hypomagnesemia (Metabolism and nutrition disorders) | 12
Hyponatremia (Metabolism and nutrition disorders) | 8
Hypophosphatemia (Metabolism and nutrition disorders) | 16
Hypotension (Vascular disorders) | 3
Insomnia (Psychiatric disorders) | 3
Lip Infection (Infections and infestations) | 1
Lipase increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 20
mucositis oral (Gastrointestinal disorders) | 8
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
nausea (Gastrointestinal disorders) | 13
Neutrophil Count Decreased (Investigations) | 18
non-cardiac chest pain (General disorders) | 1
pain (General disorders) | 6
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 5
Pancreatitis (Gastrointestinal disorders) | 1
Paresthesia (Nervous system disorders) | 1
Peripheral Motor Neuropathy (Nervous system disorders) | 3
Platelet count decreased (Investigations) | 20
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 1
prostate infection (Infections and infestations) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash Acneiform (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 10
Rectal Hemorrhage (Gastrointestinal disorders) | 1
Sinus Tachycardia (Cardiac disorders) | 1
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1
Treatment Related Secondary Malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tremor (Nervous system disorders) | 1
Urinary tract infection (Infections and infestations) | 2
Vaginal hemorrhage (Reproductive system and breast disorders) | 1
vomiting (Gastrointestinal disorders) | 10
weight loss (Investigations) | 5
White Blood Cell Decreased (Investigations) | 18
wound dehiscence (Injury, poisoning and procedural complications) | 3
wound infection (Infections and infestations) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-15): https://cdn.clinicaltrials.gov/large-docs/19/NCT02050919/Prot_SAP_000.pdf